CLINICAL TRIAL: NCT01432990
Title: Robotic Gait Training VS. Conventional Physical Therapy in Spinal Cord Injury Patients.
Brief Title: Robotic Gait Training VS.Conventional Rehabilitation in SCI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prasat Neurological Institute (Other Government)
Collaborators: Mahidol University (Other)
Responsible Party: Principal Investigator, Ratanapat Chanubol, Dr., Prasat Neurological Institute
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SCIstemcell
Record Dates: First submitted 2011-09-10; First posted 2011-09-13 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Spinal Cord Injury
Keywords: SCI; gait; rehabilitation; robotic
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- robotic gait training (Experimental): conventional physical therapy plus robot gait training program for SCI patients.
  Interventions: Device: Robot gait training
- control (No Intervention): Conventional physical therapy program for 60 minute per day for 5 working day per week.
  Interventions: Other: control

INTERVENTIONS:
Device: Robot gait training — Robotic gait training for 20 minute include preparing and rest time for 10 minute plus conventional physical therapy program for 30 minute, totally 60 minute per day for 5 working day per week.
  Other Names: Gait trainer GT1
  Arms: robotic gait training
Other: control — Conventional physical therapy program for 60 minute per day for 5 working day per week.
  Arms: control

SUMMARY:
Until now, there's still no any strong evidence supported "which is the best way to restoration walking ability" in spinal cord injury. Most of the evidence suggest that, there is somehow better after gait rehabilitation for ASIA classification C and D but not improved walking ability for ASIA classification A and B. There is an RCT showed the evidence of repetitive locomotor training and physiotherapy could be improved walking and basic activities of daily living after stroke, these might be also really effect in SCI patients.

DETAILED DESCRIPTION:
This study aim to study the effectiveness of conventional rehabilitation compare with robotic gait training machine in subacute SCI patients.

ELIGIBILITY:
Inclusion Criteria:

* Subacute spinal cord injury ( C5-T12 level) patients.
* ASIA classification C and D.
* No previous joint contracture.
* No severely active medical condition.
* Can easily communicate with no obvious cognitive impairment.
* Given signed inform consent.

Exclusion Criteria:

* Previous injury or other neurological condition that related to neurodeficit in key muscles.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Wernig scale | 4 weeks.
  Walking ability classification in spinal cord injury patients.
Barthel index | 4 weeks.
  Measure activity of daily living

SECONDARY OUTCOMES:
Repas | 4 weeks.
  Spasticity measurement
Manual muscle testing | 4 weeks
  Measure muscle power in each key muscle according to ASIA classification.
10 meter walking test | 4 weeks.
  If patients can walk, measure speed of walking with step length.
6 minute walking test | 4 weeks
  If patient can walk, measure endurance.

CONTACTS AND LOCATIONS:
Overall Officials: Ratanapat Chanubol, MD., Principal Investigator — PM&R department, Prasat Neurological Institute, Bangkok, Thailand. 10400
Locations (1):
- Ratanapat Chanubol, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Schwartz I, Sajina A, Neeb M, Fisher I, Katz-Luerer M, Meiner Z. Locomotor training using a robotic device in patients with subacute spinal cord injury. Spinal Cord. 2011 Oct;49(10):1062-7. doi: 10.1038/sc.2011.59. Epub 2011 May 31. PMID 21625239
- [Result] Pohl M, Werner C, Holzgraefe M, Kroczek G, Mehrholz J, Wingendorf I, Hoolig G, Koch R, Hesse S. Repetitive locomotor training and physiotherapy improve walking and basic activities of daily living after stroke: a single-blind, randomized multicentre trial (DEutsche GAngtrainerStudie, DEGAS). Clin Rehabil. 2007 Jan;21(1):17-27. doi: 10.1177/0269215506071281. PMID 17213237
- [Result] Tefertiller C, Pharo B, Evans N, Winchester P. Efficacy of rehabilitation robotics for walking training in neurological disorders: a review. J Rehabil Res Dev. 2011;48(4):387-416. doi: 10.1682/jrrd.2010.04.0055. PMID 21674390
- [Result] Taylor-Schroeder S, LaBarbera J, McDowell S, Zanca JM, Natale A, Mumma S, Gassaway J, Backus D. The SCIRehab project: treatment time spent in SCI rehabilitation. Physical therapy treatment time during inpatient spinal cord injury rehabilitation. J Spinal Cord Med. 2011;34(2):149-61. doi: 10.1179/107902611X12971826988057. PMID 21675354